CLINICAL TRIAL: NCT01221701
Title: Treatment of Depression in Mothers in Home Visitation
Acronym: MIDIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH073867 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Depressive Disorder in Mothers
Keywords: depression; psychological treatments; Cognitive Behavioral Therapy; child social/emotional functioning; parenting; home visitation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In-Home Cognitive Behavioral Therapy (Experimental): Mothers will receive 15 weekly sessions of IH-CBT plus one booster session scheduled 1 month later.
  Interventions: Behavioral: In-Home Cognitive Behavioral Psychology
- typical home visitation (No Intervention): Standard of care in home visitation in which mothers can receive treatment in the community if they choose.

INTERVENTIONS:
Behavioral: In-Home Cognitive Behavioral Psychology — Adapted form of CBT that is delivered in the home setting, uniquely designed for young, low income new mothers, and is explicitly integrated with home visitation. IH-CBT is delivered by a masters level therapist. It consists of 15 weekly sessions and 1 booster session provided 1 month after the 15th session.
  Other Names: IH-CBT
  Arms: In-Home Cognitive Behavioral Therapy

SUMMARY:
This study develops and contrasts In-Home Cognitive Behavioral Therapy (IH-CBT), an adapted evidence-based treatment for depressed mothers participating in home visitation, with typical home visitation in which treatment may be obtained in the community. Mothers will be identified using a two step process consisting of administration of a screen and subsequent diagnosis of Major Depressive Disorder. The will then be randomized into the treatment and control conditions. A comprehensive assessment of depression and related areas of functioning will be administered at pre-treatment, post-treatment, and 3 month follow-up. It is hypothesized that IH-CBT will lead to broad and durable gains in mood and social support relative to those in typical home visitation.

DETAILED DESCRIPTION:
This study involves the development and preliminarily testing of In-Home Cognitive Behavioral Therapy (IH-CBT), a psychological treatment grounded in the cognitive model but adapted for administration in conjunction with home visitation. IH-CBT is designed to (1) use the techniques and approaches of CBT which have received strong empirical support, (2) be implemented in the home setting, (3) meet the needs of young postpartum mothers in their first year of home visitation, and (4) be seamlessly integrated with home visitation to maximize the likelihood of recovery from depression, prevent relapse, and increase of the benefits of home visitation. IH-CBT will be delivered by trained therapist who will provide 15 treatment sessions followed by a 1 month booster session. A small-scale randomized clinical trial will be conducted contrasting IH-CBT delivered in conjunction with home visitation and home visitation alone ("typical home visitation"-THV). Mothers in the THV condition will be able to obtain treatment in the community if they choose.

Mothers will be identified based on obtaining a score of ≥12 on the Edinburgh Perinatal Depression Screen administered by home visitors at 3 months postpartum. Final eligibility will be determined based on subsequently obtaining a diagnosis of Major Depressive Disorder (MDD) using the SCID. A comprehensive assessment of depression, other psychiatric symptoms, social support and network, and parenting and child adjustment will be administered at pre-treatment, post-treatment, and 3 month follow-up. Ratings of MDD at post-treatment and follow-up will be conducted by clinicians blind to condition.

The following hypotheses will be tested:

Hypothesis 1. Mothers in IH-CBT will report greater reductions in self-reported and clinician-rated depression at post-treatment and follow up relative to THV.

Hypothesis 2. Mothers in IH-CBT will report improvements in overall functioning, social support, social network, and general psychiatric symptomatology at post-treatment and follow up relative to IH-CBT.

Hypothesis 3. Mothers who recover from depression at post-treatment will report improvements in parenting and child adjustment relative to those who do not recover.

ELIGIBILITY:
Inclusion Criteria:

* first-time mother participating in home visitation program
* enrolled in home visitation program for at least 2 months
* 16 years of age or older
* score of 12 or higher on Edinburgh Perinatal Depression Screen at 3 months postpartum
* diagnosis of Major Depressive Disorder using the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders
* English speaking

Exclusion Criteria:

* lifetime history of bipolar disorder, schizophrenia, mental retardation, organic brain syndrome, antisocial personality disorder
* history of psychosis
* current substance dependence
* current antidepressant use or other mood altering medications and/or current involvement in psychotherapy

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 2006-10; Primary Completion 2010-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
maternal depression | 8 months
  Maternal depression as measured by self-report, clinician rating based on semi-structured interview, and psychiatric diagnosis based on semi-structured interview.

SECONDARY OUTCOMES:
parenting and child social/emotional functioning | 8 months
  Maternal report of parenting stress, observation of parenting behaviors, and maternal report of child social/emotional functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Robert T. Ammerman, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Ammerman RT, Putnam FW, Bosse NR, Teeters AR, Van Ginkel JB. Maternal Depression in Home Visitation: A Systematic Review. Aggress Violent Behav. 2010 May;15(3):191-200. doi: 10.1016/j.avb.2009.12.002. PMID 20401324
- [Background] Ammerman RT, Putnam FW, Stevens J, Bosse NR, Short JA, Bodley AL, Van Ginkel JB. An open trial of in-home CBT for depressed mothers in home visitation. Matern Child Health J. 2011 Nov;15(8):1333-41. doi: 10.1007/s10995-010-0691-7. PMID 20936338